CLINICAL TRIAL: NCT04002999
Title: Precision Orthodontics: Customized Versus Conventional Orthodontic Bracket Prescriptions - A Randomized Controlled Clinical Trial
Brief Title: Precision Orthodontics: Virtual Treatment Planning for Orthodontic Braces
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Harvard School of Dental Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 18-0615
Record Dates: First submitted 2019-06-27; First posted 2019-07-01 (Actual); Last update posted 2020-02-12 (Actual); Status verified 2019-04

CONDITIONS: Malocclusion; Malocclusion, Angle's Class
Keywords: 3D printing; Virtual treatment planning
MeSH Terms: conditions — Malocclusion

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Ceramic braces, directly placed (Active Comparator): Patients in this group will be treated with directly-bonded traditional tooth-colored ceramic brackets
  Interventions: Device: Stock bracket, no tray
- Ceramic braces, indirectly placed (Experimental): Patients will be treated with the same brackets from treatment group 1 but using the indirect bonding technique
  Interventions: Device: Stock ceramic bracket + 3D printed tray
- 3D printed customized ceramic braces (Experimental): Patients will be treated using indirectly bonded 3D-printed ceramic (tooth-closed) brackets
  Interventions: Device: 3D printed ceramic bracket and tray

INTERVENTIONS:
Device: 3D printed ceramic bracket and tray — The 3D ceramic bracket being investigated is the only available customized ceramic bracket. This will be a first for the orthodontic speciality. This will also be the first and only customized bracket system that includes customization of the bracket base. This helps in the control of first order orthodontic movements and allows brackets to be bonded on any labial surface of the tooth while maintaining an ideal prescription. As 3D printing is not limited by the mold-ejection in CIM, [24] the bracket system being tested here has the potential to achieve a more accurate slot dimension.
  Arms: 3D printed customized ceramic braces
Device: Stock ceramic bracket + 3D printed tray — Traditionally, indirect bonding, starts with creating a mold of all the teeth as an exact replica of the mouth of the patient. From there, in the lab, the orthodontist positions each bracket precisely where it should go on each tooth and then creates a custom tray that allows transfer of the brackets from the lab model to the patient's teeth. By taking the time to place the brackets in a proper position on the lab model, orthodontists eliminate the inaccurate process of placing orthodontic brackets directly on the teeth. It theoretically also takes less chairside time and is more comfortable for the patient. It is however more technique sensitive. In this study, indirect bonding setup will be done virtually using commonly-available orthodontic software. The trays/jigs will then be 3-D printed
  Arms: Ceramic braces, indirectly placed
Device: Stock bracket, no tray — Direct bonding is the traditional way of placing orthodontic brackets, in which orthodontists clinically eyeball the tooth and place the bracket where they deem most appropriate
  Arms: Ceramic braces, directly placed

SUMMARY:
The investigators are evaluating the effectiveness of custom-made 3D-printed ceramic (tooth-colored) brackets (braces) compared to conventional tooth-colored brackets (braces).

Participants will be expected to come in for regularly scheduled appointments. They will be treated with tooth-colored braces and will need to come in every 4-6 weeks and will be randomly assigned to one of three groups. "Randomly" means by chance, like a coin toss. Neither participants nor the researchers may choose group assignments. Group 1 patients will have tooth-colored braces placed directly on each tooth by the clinician. Group 2 patients will have the braces placed on the teeth by using trays to fit them on. Group 3 patients will have customized 3D printed tooth-colored braces placed on their teeth, using trays to fit them on. If a participant is selected to be part of group 3, it may take up to two additional weeks for these 3D brackets to be printed and shipped and so this might delay treatment onset. Information on gender, age, and medical history of participants will also be obtained from the electronic health record.

DETAILED DESCRIPTION:
Teeth and orthodontic treatment plans are very unique to the specific patient, yet standard orthodontic braces are currently "one-size fits all". In the early 20th century, orthodontics was practiced using non-programmed brackets. First, second and third order bends had to be incorporated into the wire in order to achieve ideal final tooth positions.

Andrews' Straight Wire Appliance (SWA) in the 1970s, however, revolutionized orthodontic care by presenting a standard set of brackets with pre-programmed prescriptions built into the appliance system [5-7]. According to Andrews, "it is far easier to control tooth movement with bracket placement than bending wires".

Andrews analyzed 120 patient cases which presented with what he described as an ideal occlusion. He documented common characteristics in regard to angulation, tip, and torque subjectively deemed to create an ideal occlusion. This allowed him to develop a bracket prescription to compensate for the disparity in the contour of the facial surfaces of teeth by increasing thickness of the bracket base. Furthermore, he introduced angulations within the bracket slot to achieve proper positioning of the roots [5, 8]. This "straight-wire appliance" (SWA) method became widely accepted in orthodontics, and numerous variations of pre-adjusted bracket systems have since been introduced. Pre-adjusted brackets, however, fail to address deviations from average tooth morphology and other treatment nuances. These are often tackled chairside by placing bends on arch wires [9-12] - bends that the SWA method was invented to prevent. Additionally, mechanical boundaries and imprecision of bracket placement can result in limitations to treatment. [13-15] All these inaccuracies may cumulate during the course of a treatment to increase treatment time, resulting in frustration and compromised results.

Technological advancements have allowed for some customization of brackets and wires in order to address limitations of conventional pre-adjusted bracket systems. Digital intra-oral scans are obtained at the onset of treatment to generate a digital study model of the dentition. Virtual models are analyzed to determine the ideal position of each tooth required for achieving stable occlusion. Those digital models also allow for bracket positioning set-up; indirect-bonding transfer jigs allow virtual positioning to be replicated intra-orally. The clinician creates a virtual design of the final occlusion and alignment using computer-assisted technology, with reverse-engineered brackets and archwires used to obtain the intended result. Bracket slots are customized to accommodate a straight wire that moves each tooth to the ideal final position as identified by the virtual setup. Virtual bracket positions are then transferred to the patient by means of indirect-bonding transfer jigs [16].

Several orthodontic systems implement some of these new technologies, [17] providing the orthodontist with a treatment package consisting of digital diagnostics, 3-dimensional (3D) digital planning, and computer-designed customized brackets and arch wires. One such system is the Insignia (ORMCO Corporation) system [18], which entered the market several years ago. Theoretically, individualized orthodontic treatment systems offer several advantages for both the patient and orthodontist, with commonly mentioned benefits including better treatment results, shorter treatment duration, and less chair time. [19] Manufacturers utilizing virtual treatment planning and customized, computer-aided fabrication of tooth supported orthodontic appliances claim to deliver superior quality and efficiency of care compared to conventional preadjusted bracket systems. To date, few studies have investigated the accuracy of these systems in achieving their virtually planned tooth positions.

A 2015 retrospective study [20] reported that a Computer-aided design/computer-aided manufacturing (CAD/CAM) orthodontic bracket system (Insignia ®) produced similar treatment outcomes compared with direct and indirect bonded appliances. The CAD/CAM group nonetheless had shorter treatment times than the direct and indirect bonded groups. To our knowledge, only one prospective randomized clinical trial (RCT) [21] has explored the advantage or otherwise of partially customized appliances with precise placement over directly or indirectly bonded stock brackets.

The above-referenced RCT [21] concluded that "compared to the non-customized system, the customized orthodontic system was not associated with any significant reduction in treatment duration, and the treatment outcomes were comparable with both systems. Treatment duration and quality were affected by the orthodontist and the severity of malocclusion at the start of treatment rather than by the orthodontic system used. Treatment with a customized appliance, such as the one used in this trial, required significantly more planning time from the orthodontist and was associated with a higher number of visits due to loose brackets." This study, however, introduced significant variability between the two test groups by using two different bonding techniques. As a result, their conclusions could be flawed. Beyond this, the customized brackets they used did not include customization of the bracket base to conform to tooth anatomy. This is important because bracket base-tooth surface discrepancies can lead to inaccuracies in the final in-out position of the tooth.

Due to recent breakthroughs in the area of 3D printing in dentistry - precisely, additive manufacturing (AM) - and the limitations of previous studies (lack of randomization/appropriate control for potential confounders), the need arises to evaluate if 3D-printed ceramic brackets offer any superiority to traditional ceramic braces.

Minimizing errors and improving accuracy are important factors not only for patient satisfaction, but also for preventing adverse effects such as root resorption that occur when unwanted tooth movements occur [22]. Different strategies have been designed for this purpose, foremost among which has been to enhance treatment outcomes by precisely planning tooth movements and positioning brackets with greater accuracy. Since the early stages of multi-bracket appliance development, it was clear that precise bracket placement is key to the success of the straight-wire concept [10]. One author stated that it is impossible to solve the problem of adapting a bracket to a patient's specific tooth and to individualize treatment goals without individualizing at least one bracket component and that new additive manufacturing (AM) options can provide the catalyst for future developments in this field [23]. Treatment with computer-designed customized brackets has the potential to personalize orthodontic care, but the benefits remain to be validated. The present randomized controlled trial aims to compare orthodontic treatment effectiveness in a customized versus non-customized ceramic orthodontic system.

2. Innovation The 3D ceramic bracket being investigated is the only available customized ceramic bracket. This will be a first for the orthodontic speciality. This will also be the first and only customized bracket system that includes customization of the bracket base. This helps in the control of first order orthodontic movements and allows brackets to be bonded on any labial surface of the tooth while maintaining an ideal prescription. As 3D printing is not limited by the mold-ejection in CIM (ceramic injection molding) [24] the bracket system being tested here has the potential to achieve a more accurate slot dimension. This is important because a critical factor affecting the expression of a bracket prescription is the accuracy of the bracket slot. Various orthodontic textbooks have defined expectations for bracket slot accuracy. In Contemporary Orthodontics, Proffitt et al. [25] stated that the precision of orthodontic bracket manufacturing should render slot dimension accuracy of at least 1 mil to ensure accurate expression of a chosen prescription. Oversized slots (due to manufacturing limitations) defeat the premise of prescription orthodontic brackets as the larger slot size does not allow for complete prescription expression [26].

3.1 Design This will be a parallel-arm randomized controlled clinical trial that involves 3 treatment groups

3.1.1 Treatment groups Treatment group 1: Patients in this group will be treated with directly-bonded traditional (stock) .018 ceramic brackets Treatment group 2: Patients will be treated with the same brackets from treatment group 1 but using the indirect bonding (IDB) technique Treatment group 3: Patients will be treated using indirectly bonded fully customized 3D-printed ceramic brackets. All participating clinicians will be trained in digital orthodontics, and the IDB technique through hands-on sessions by orthodontists who are experienced in the use of IDB and digital set up.

Direct bonding is the traditional way of placing orthodontic brackets, in which orthodontists clinically eyeball the tooth and place the bracket where they deem most appropriate. Traditionally, indirect bonding, starts with creating a mold of all the teeth as an exact replica of the mouth of the patient. From there, in the lab, the orthodontist positions each bracket precisely where it should go on each tooth and then creates a custom tray that allows transfer of the brackets from the lab model to the patient's teeth. By taking the time to place the brackets in a proper position on the lab model, orthodontists eliminate the inaccurate process of placing orthodontic brackets directly on the teeth. It theoretically also takes less chairside time and is more comfortable for the patient. It is however more technique sensitive. In this study, indirect bonding setup will be done virtually using commonly-available orthodontic software. The trays/jigs will then be 3-D printed.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects over the age of 10 years and below 65;
* Eruption of all permanent teeth excluding second and third molars;
* Non-extraction treatment;
* Maximum of 7mm of crowding/spacing;
* No more than 45 degrees of rotations

Exclusion Criteria:

* Presence of systemic diseases, cleft lip and palate, craniofacial anomalies, syndromes affecting bone or teeth, impacted teeth (excluding 3rd molars); congenitally missing teeth, and tumors of the parathyroid gland;
* The presence of bridges or implants;
* Significant (> moderate) periodontal disease, intake of drugs affecting tooth movement or bone formation (chronic use of Non-Steroidal Anti-Inflammatory Drugs, bisphosphonates, levothyroxine, or teriparatide drug class), pregnancy; and
* Cases requiring tooth extractions

Ages: 11 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 51 (Estimated)
Dates: Start 2019-08-30 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
Quality of first stage of orthodontic finish: Objective Grading System (OGS) | 12months
  A number of measures have been developed to determine the quality of orthodontic treatment. The Objective Grading System (OGS), [27] developed by the American Board of Orthodontics (ABO) in 1994, was designed to establish a uniform and objective evaluation of cases

CONTACTS AND LOCATIONS:
Locations (1):
- Harvard Dental Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No